CLINICAL TRIAL: NCT05514379
Title: Disorders of Gait, Postural Stability and Cognition in Parkinson's Disease: Presymptomatic Detection and Targeted Rehabilitation
Brief Title: Effect of Cognitive Training on Gait in Parkinson's Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: General University Hospital, Prague (Other)
Collaborators: Charles University, Czech Republic (Other)
Responsible Party: Principal Investigator, Evžen Růžička, Prof. Evzen Ruzicka, MD, DSc., General University Hospital, Prague
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NU20-04-00327
Record Dates: First submitted 2022-08-15; First posted 2022-08-24 (Actual); Last update posted 2023-09-14 (Actual); Status verified 2023-09

CONDITIONS: Parkinson Disease
Keywords: Parkinson Disease; Cognitive training; Gait
MeSH Terms: conditions — Parkinson Disease | interventions — Cognitive Training

STUDY DESIGN:
Intervention Model Description: Prticipants are randomly assigned to either the experimental or the control group.
Who Masked: Participant, Investigator
Masking Description: Participants are blinded to study hypothesis. Investigators are blinded to treatment group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group cognitive training (Experimental): The experimental group will undergo 60 minutes long cognitive training group sessions twice a week for 12 weeks focused on executive function, attention and working memory.
  Interventions: Behavioral: cognitive training
- Home-based cognitive training (Active Comparator): The control group will perform executive function, attention and working memory training similar to the experimental group but at home as instructed by their therapist using specialized software for cognitive training (Rehacom). This training will be dose matched to the experimental group, i.e. it will be performed four times a week for 30 minutes for 12 weeks. In this group, therapists will only provide coaching once a month.
  Interventions: Behavioral: cognitive training

INTERVENTIONS:
Behavioral: cognitive training — Cognitive training focused on executive function, attention and working memory delivered either by the therapist in a group setting (experimental group) or by a specialized software for cognitive training (Rehacom) at home.

SUMMARY:
Physiotherapy and targeted rehabilitation are routinely performed in order to influence disorders of posture, gait and stability in Parkinson´s disease (PD), but their effects have been controversial (Keus et al. 2014; Walton wt al. 2014). Recently, several studies suggested that cognitive training can improve gait in patients with PD (Peterson et al. 2016, Heremans et al. 2013), similar to the effects seen in the elderly (Yogev-Seligmann et al. 2008; Amboni et al. 2013). Specific training programs including dual tasking with automatic verbal series, counting etc. have led to increased walking speed and improved stepping cadence, length, and duration in patients with dementia (Schwenk et al. 2010). However, since in advanced PD patients dual-task gait training has to be supervised by therapists, it is not a suitable type of therapy to be performed at home. Therefore, this study aims to verify and extend the encouraging results of the single study which showed a positive effect of cognitive function training on gait in PD (Milman et al. 2014) by exploring this effect in advanced PD patients, by assessing the effect on gait using more targeted clinical and instrumental evaluation, and by comparing two modes of therapy delivery, group and computer-based.

DETAILED DESCRIPTION:
* Background: In a pilot study, Milman et al. 2014 showed that computer-based cognitive training focusing on executive function and attention performed at home might improve selected gait parameters in early patients with Parkinson´s disease (PD).
* Goal 1: To explore this effect in advanced PD patients
* Hypothesis 1: Effect of cognitive training focusing on executive function and attention will be detected also in advanced PD patients and this effect will be larger as compared to the results published by Milman et al. 2014.
* Goal 2: To verify the results published by Milman et al. 2014 using more targeted clinical and instrumental gait assessment, including dual-task gait evaluation as well as instrumental testing of turn fluency (Bertoli et al. 2019).
* Hypothesis 2: The results published by Milman et al. 2014 will be confirmed and an effect on dual-task gait and turn fluency will be shown.
* Goal 3: To explore the role of the form of therapy setting, i.e. whether group setting might increase the effect of cognitive training on gait as compared to individual cognitive training at home. Such results have been shown in the case of a physiotherapy intervention by King et al. 2015.
* Hypothesis 3: The effect of group cognitive training on gait will be larger as compared to individual dose-matched, computer-based cognitive training performed at home. However, it remains to be determined whether the effect size difference between the two groups will outweigh the advantages of tele-rehabilitation.
* Design: Randomised-controlled trial
* Interventions: experimental group: group cognitive training focusing on executive function and attention; control group: computer-based cognitive training focusing on executive function and attention performed at home. Intervention in both groups will be dose-matched (experimental: 60 mins, 2x/week, 12 weeks; control: 30 mins, 4x/week, 12 weeks)
* Follow-up: at 1 and 3 months time points.
* Power analysis results: at least 38 patients.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of Parkinson´s disease (PD)
* PD duration ≥8 years
* mild cognitive impairment
* stable medication
* presence of freezing of gait according to the FoG-Q AND/OR Rapid Turns Test

Exclusion Criteria:

* dementia
* deep brain stimulation, pump therapy with Duodopa or Apomorphine
* severe fluctuations with ON state duration for less than 2 hours
* dopa dysregulation syndrome
* impulse control disorder
* untreated depression
* benzodiazepines except for single dose at night
* non-compliance
* inability to walk without support
* significant co-morbidities likely to affect gait, e.g., acute illness, orthopedic disease, significant visual problems, or a clinical history of stroke
* involvement in other treatment trials
* not meeting inclusion criteria

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2023-10 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline instrumental assessment of turn fluency during rapid turns at 12 weeks | Baseline and 12 weeks
  see Bertoli et al. 2019 for a detailed description; G-Walk instrumental gait assessment will be used
Change from Baseline Timed Up and Go Test: dual-task performance at 12 weeks | Baseline and 12 weeks
  Patient is asked to perform TUG while subtracting 3 from a random number between 51-100; G-Walk instrumental gait assessment will be used

SECONDARY OUTCOMES:
Timed Up and Go Test: single-task performance | Baseline, 12 weeks, 1 month follow-up, 3 months follow-up
  G-Walk instrumental gait assessment will be used
10-meter walking test: single-task performance | Baseline, 12 weeks, 1 month follow-up, 3 months follow-up
  G-Walk instrumental gait assessment will be used
10-meter walking test: dual-task performance | Baseline, 12 weeks, 1 month follow-up, 3 months follow-up
  Patient is asked to perform 10MWT while subtracting 3 from a random number between 51-100; G-Walk instrumental gait assessment will be used
Number of steps/day | 5 days monitoring at baseline and 12 weeks
  Assessed using Fitbit activity trackers
The Montreal Cognitive Assessment (MoCA), Total score | Baseline, 12 weeks, 3 months follow-up
  Global cognition screening
Trail Making Test A (TMT A), Total score (in seconds) | Baseline, 12 weeks, 1 month follow-up, 3 months follow-up
  Assessing of attention distribution.
The Victoria Version of Stroop Test (VST): Dot Time Score (in seconds) Neutral Word Time Score (in seconds) The Victoria Version of Stroop Test (VST): Dot Time Score (in seconds) Neutral Word Time Score (in seconds) | Baseline, 12 weeks, 1 month follow-up, 3 months follow-up
  Assessing of focused visual attention
The Victoria Version of Stroop Test (VST): Color Word Time Score (in seconds) Error score on VST Color Word Task, Total score | Baseline, 12 weeks, 1 month follow-up, 3 months follow-up
  Assessing of executive functions - inhibition
Tower of London, Total score | Baseline, 12 weeks, 1 month follow-up, 3 months follow-up
  Assessing of executive functions - problem solving
Depression, Anxiety and Stress Scale (DASS 21) | Baseline, 12 weeks, 1 month follow-up, 3 months follow-up
  Self-assessment scale of depression, anxiety and stress. Patient fills it at home.
Falls Efficacy Scale-International | Baseline, 12 weeks, 1 month follow-up, 3 months follow-up
  Fear of falls assessment
Number of falls | Baseline, 12 weeks, 1 month follow-up, 3 months follow-up
  Diary based quantification of the number of falls
Change from post-intervention instrumental assessment of turn fluency during rapid turns at 1 month follow-up | 12 weeks and 1 month follow-up
  see Bertoli et al. 2019 for a detailed description; G-Walk instrumental gait assessment will be used
Change from post-intervention instrumental assessment of turn fluency during rapid turns at 3 months follow-up | 12 weeks and 3 months follow-up
  see Bertoli et al. 2019 for a detailed description; G-Walk instrumental gait assessment will be used
Change from post-intervention Timed Up and Go Test: dual-task performance at 1 month follow-up | 12 weeks and 1 month follow-up
  Patient is asked to perform TUG while subtracting 3 from a random number between 51-100; G-Walk instrumental gait assessment will be used
Change from post-intervention Timed Up and Go Test: dual-task performance at 3 months follow-up | 12 weeks and 3 months follow-up
  Patient is asked to perform TUG while subtracting 3 from a random number between 51-100; G-Walk instrumental gait assessment will be used

OTHER OUTCOMES:
Counting: number of (correct) answers per second | Baseline, 12 weeks, 1 month follow-up, 3 months follow-up
  Patient is asked to subtract 3 from a random number between 51-100 while seated. This assessment is used as a reference value for TUG-DT and 10MWT-DT
MDS-Unified Parkinson's Disease Rating Scale | Baseline, 12 weeks, 1 month follow-up, 3 months follow-up
  Scale evaluating various aspects of Parkinson's disease including non-motor and motor experiences of daily living and motor complications.
Freezing of Gait Questionnaire | Baseline, 12 weeks, 1 month follow-up, 3 months follow-up
  Subjective evaluation of freezing of gait
Quantitative MRI metrics | Baseline
  Volumetric parameters
Quantitative MRI metrics | Baseline
  Vascular white matter lesional volume
Quantitative MRI metrics | Baseline
  Resting functional connectivity
Auditory Verbal Learning Test (AVLT): T1 (Try) T2 T3 T4 T5 T1-5 Total score Interfence, Total score T6, Total score Delayed recall, Total score Recognition, Correct answers total score, False answers total score | Baseline, 12 weeks, 1 month follow-up, 3 months follow-up
  Assessing of auditory memory, memory capacity, ability to learn, delayed recall, recognition
Phonemic Verbal Fluency FAS, letters: K, P, S Letter K, Total score Letter P, Total Score Letter S, Total score Letters K, P, S, Total score | Baseline, 12 weeks, 1 month follow-up, 3 months follow-up
  Assessing of executive functions - initation, maintenance, stop and end the activity
Semantic Fluency, category: Animals, Total score | Baseline, 12 weeks, 1 month follow-up, 3 months follow-up
  Assessing of phatic functions.
Trail Making Test B (TMT B): Total score (in seconds), Number of errors | Baseline, 12 weeks, 1 month follow-up, 3 months follow-up
  Assessing of executive functions - cognitive flexibility.
Digit Span Forward, Wechsler Adult Intelligence Scale-Revised, Total score Digit Span Forward, Wechsler Adult Intelligence Scale-Revised, Total score | Baseline, 12 weeks, 1 month follow-up, 3 months follow-up
  Assessing of focused auditory attention.
Digit Span Backward, Wechsler Adult Intelligence Scale-Revised, Total score | Baseline, 12 weeks, 1 month follow-up, 3 months follow-up
  Working memory capacity measurement.
Digit Symbol, Wechsler Adult Intelligence Scale-Revised, Total score | Baseline, 12 weeks, 1 month follow-up, 3 months follow-up
  Assessing of divided attention and working memory.
Grooved Pegboard, Left. | Baseline, 12 weeks, 1 month follow-up, 3 months follow-up
  Assessing of visual-motor coordination. The Grooved Pegboard is a manipulative dexterity test consisting of 25 holes with randomly positioned slots. Pegs with a key along one side must be rotated to match the hole before they can be inserted.
The Parkinson´s Disease Questionnaire (PDQ-39) | Baseline, 12 weeks, 1 month follow-up, 3 months follow-up
  Self-assessment quality of life scale for patients with Parkinson's disease. Patient fills it at home.
Grooved Pegboard, Right. | Baseline, 12 weeks, 1 month follow-up, 3 months follow-up
  Assessing of visual-motor coordination. The Grooved Pegboard is a manipulative dexterity test consisting of 25 holes with randomly positioned slots. Pegs with a key along one side must be rotated to match the hole before they can be inserted.
Exploratory assessment of relationship between clinical effects of cognitive training and blood signature of polymorphisms in PD-related genes | Baseline
  Custom genetic panel (SureSelect, Agilent) for mutational analysis of 177 genes (including APOE, MAPT, GBA LRRK2, etc.)

CONTACTS AND LOCATIONS:
Overall Officials: Evzen Ruzicka, Prof., Principal Investigator — General University Hospital, Prague
Locations (1):
- General University Hospital in Prague, Prague, Czechia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Milman U, Atias H, Weiss A, Mirelman A, Hausdorff JM. Can cognitive remediation improve mobility in patients with Parkinson's disease? Findings from a 12 week pilot study. J Parkinsons Dis. 2014;4(1):37-44. doi: 10.3233/JPD-130321. PMID 24322063
- [Background] Yogev-Seligmann G, Hausdorff JM, Giladi N. The role of executive function and attention in gait. Mov Disord. 2008 Feb 15;23(3):329-42; quiz 472. doi: 10.1002/mds.21720. PMID 18058946
- [Background] Amboni M, Barone P, Hausdorff JM. Cognitive contributions to gait and falls: evidence and implications. Mov Disord. 2013 Sep 15;28(11):1520-33. doi: 10.1002/mds.25674. PMID 24132840
- [Background] Keus SHJ MM, Graziano M, et al. European Physiotherapy Guideline for Parkinson´s Disease. the Netherlands: KNGF/ParkinsonNet,2014.
- [Background] Walton CC, Shine JM, Mowszowski L, Naismith SL, Lewis SJ. Freezing of gait in Parkinson's disease: current treatments and the potential role for cognitive training. Restor Neurol Neurosci. 2014;32(3):411-22. doi: 10.3233/RNN-130370. PMID 24531294
- [Background] Peterson DS, King LA, Cohen RG, Horak FB. Cognitive Contributions to Freezing of Gait in Parkinson Disease: Implications for Physical Rehabilitation. Phys Ther. 2016 May;96(5):659-70. doi: 10.2522/ptj.20140603. Epub 2015 Sep 17. PMID 26381808
- [Background] Heremans E, Nieuwboer A, Spildooren J, Vandenbossche J, Deroost N, Soetens E, Kerckhofs E, Vercruysse S. Cognitive aspects of freezing of gait in Parkinson's disease: a challenge for rehabilitation. J Neural Transm (Vienna). 2013 Apr;120(4):543-57. doi: 10.1007/s00702-012-0964-y. Epub 2013 Jan 18. PMID 23328947
- [Background] Schwenk M, Zieschang T, Oster P, Hauer K. Dual-task performances can be improved in patients with dementia: a randomized controlled trial. Neurology. 2010 Jun 15;74(24):1961-8. doi: 10.1212/WNL.0b013e3181e39696. Epub 2010 May 5. PMID 20445152
- [Background] Bertoli M, Croce UD, Cereatti A, Mancini M. Objective measures to investigate turning impairments and freezing of gait in people with Parkinson's disease. Gait Posture. 2019 Oct;74:187-193. doi: 10.1016/j.gaitpost.2019.09.001. Epub 2019 Sep 5. PMID 31539800
- [Background] King LA, Wilhelm J, Chen Y, Blehm R, Nutt J, Chen Z, Serdar A, Horak FB. Effects of Group, Individual, and Home Exercise in Persons With Parkinson Disease: A Randomized Clinical Trial. J Neurol Phys Ther. 2015 Oct;39(4):204-12. doi: 10.1097/NPT.0000000000000101. PMID 26308937